CLINICAL TRIAL: NCT00252967
Title: Atorvastatin Therapy for the Prevention of Atrial Fibrillation (SToP-AF)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient power to show therapy difference at interim analysis.
Sponsor: Emory University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Samuel C. Dudley, Jr., MD, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB00024771; 1137-2004 (Other: Other)
Record Dates: First submitted 2005-11-14; First posted 2005-11-15 (Estimated); Results first posted 2014-09-03 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-08

CONDITIONS: Atrial Fibrillation; Inflammation
Keywords: Reactive Oxgen Speers; Atrial Fibrillation; Oxidative Stress; Inflammation
MeSH Terms: conditions — Atrial Fibrillation; Inflammation | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo taken daily
  Interventions: Drug: Placebo
- Atorvastatin (Experimental): Atorvastatin at a dose of 80 mg daily
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — 80 mg of Atorvastatin
  Arms: Atorvastatin
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to test whether the drug, atorvastatin, will be able to reduce the rate of return of the abnormal beats after using cardioversion. Atorvastatin is a drug approved by the Food and Drug Administration (FDA) for the treatment of high cholesterol but is not approved for preventing abnormal heartbeats. In addition to lowering cholesterol, the drug reduces inflammation. Inflammation seems to help cause atrial fibrillation, a certain type of abnormal heartbeat. In animals, atorvastatin reduces the risk of this type of abnormal beats, and preliminary data in humans supports an effect of atorvastatin and other similar drugs that have the same action on reducing the risk of this type of abnormal beats. We, the researchers at Emory University, would like to learn if this drug could prevent the return of these abnormal heartbeats.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) and its related disorder, atrial flutter (AFlut), are common abnormal heartbeats. Because they are similar and AFlut is rare compared to AF, they are usually treated similarly and discussed as one disorder. AF is an extremely common arrhythmia affecting more that 5% of the population over 65 years of age. It is an independent risk factor for death. AF is considered a progressive disease increasing in prevalence with age and converting from paroxysmal to permanent within a single individual. The projected lifetime risk of AF is 1 in 4 for men. AF occurs when there is an electrical short circuit in the top parts of the heart (atria). This causes the atria to beat at >300 times per min in an irregular and ineffective manor. This has two consequences. The blood tends to pool in the atria allowing for clotting. Second, the bottom parts of the heart (ventricles) beat too rapidly in response to impulses arising in the atria. The rapid ventricular contraction without adequate filling time results in a reduced ejection of blood. This can cause heart failure symptoms such as shortness of breath and reduced blood flow to organs resulting in lightheadedness or collapse.

One logical therapy to correct the defects arising from AF is return the abnormal heartbeats back to the normal rhythm. This can be done with electrical shock therapy (cardioversion) or by drugs called antiarrhythmic agents. Often, they are used together. While its stands to reason that using these techniques to restore rhythm to normal would be beneficial, clinical trials show that leaving patients in AF and thinning the blood to prevent blood clots is equally efficacious to trying to restore normal beating (sinus rhythm). The common explanations for this are that AF returns rapidly despite antiarrhythmic drugs and that antiarrhythmic drugs can make worse abnormal heart beats, a phenomenon known as proarrhythmia.

Based on the lack of efficacy of current therapies and similarities between risk factors for atherosclerosis (hardening of the arteries) and AF, we began to investigate whether oxidative stress, a mechanism similar to inflammation thought to be responsible for atherosclerosis, might be playing a role in causing AF. We studied this in pigs first and found that when we put pigs into AF, they had a large increase in oxidative stress markers. Then, we made a mouse that had too much oxidative stress in the heart, and this mouse developed AF. Based on this and other data in humans, we hypothesized that oxidative stress can cause AF.

Atorvastatin is a cholesterol lowering medication that works by blocking production of cholesterol at an early stage. This has the effect of preventing the synthesis of molecules required to assemble the most common enzymatic source of oxidative stress, the NADPH oxidase. Therefore, atorvastatin decreases oxidative stress in addition to reducing cholesterol, and if our hypothesis is correct, atorvastatin should reduce the incidence of AF.

In this study we chose to look at patients undergoing cardioversion. This is because this group has a high likelihood of recurrence of AF and would benefit most by an effective drug. Once the decision is made to have the patient undergo cardioversion, we will approach the patient about enrolling in this trial. The only change in their medical therapy will be the addition of the study drug. The study requires no other alterations to the standard of care. If patients agree to participate, then they will be started on the study drug and followed for recurrence of AF by a variety of surface electrocardiogram techniques. All of which are noninvasive. To insure the medicine is not causing side effects, examinations and blood tests will be done, and to study whether the drug actually affects oxidative stress, blood will be analyzed. The subjects participation ends when AF recurs or after 1 year. This will be a double blind, placebo controlled trial and will be analyzed on an intention to treat basis.

The risks of this study to the patient are likely to be small compared to the potential benefit of reduced AF burden. Based on a previous trial using the same dose of study medication, the risks of all study drug related adverse events is likely to be <3%. All of these are expected to be reversible with discontinuation of the drug.

The significance of this research is that currently treatments to address AF are less than optimal. Antiarrhythmic drugs are variably effective and are associated with potentially lethal proarrhythmic side effects. The common treatment to prevent strokes in subjects with AF is chronic warfarin administration, but warfarin therapy requires frequent monitoring and adjustment of dose and is associated with bleeding complications. This research may provide the first new therapeutic strategy in many years for AF and the most serious consequence of AF, stroke.

ELIGIBILITY:
Inclusion Criteria:

* > or = 18 years of age
* Clinical diagnosis-abnormal heart beat known as atrial fibrillation/flutter (ECG documentation)
* Able to swallow pill form of drug

Exclusion Criteria:

* < 18 years of age
* enrollment in another ongoing trial
* paroxysmal atrial fibrillation
* hemodynamic instability
* atrial fibrillation ablation within 6 months of enrollment
* a contraindication for anticoagulation
* severe valvular heart disease
* presence of single lead implantable cardioverter defibrillator
* unstable angina
* New York Heart Association (NYHA) Class IV heart failure
* hyperthyroidism
* uncontrolled hypertension (blood pressure > 180/100 at rest) on medications
* an illness that would limit life expectancy to less than 1 year
* use of statins within the previous 30 days
* significant coronary artery disease or lipid abnormalities necessitating statin therapy
* implanted devices for active management of arrhythmias by pacing or defibrillation
* lack of access to a telephone
* illicit drug use
* alcohol abuse
* hypersensitivity to atorvastatin by history
* pregnancy
* sexually active female subjects not on contraception or surgically sterilized
* nursing mothers
* chronic liver disease or abnormal liver function (elevated transaminases 1.5 times the upper limit of normal [ULN] of laboratory reference range)
* severe renal disease (creatinine > 200 mmol/L)
* inflammatory muscle disease or creatine kinase (CK) > 3 times ULN
* concurrent treatment with cyclosporine, fibrates, or high-dose niacin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2005-10; Primary Completion 2008-11 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel D. Dudley, Jr., MD, PhD, Principal Investigator — US Department of Veterans Affairs
Locations (3):
- United States (3):
  - Veteran Administration Medical Center/Emory University, Atlanta, Georgia
  - Crawford Long Hospital, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia

REFERENCES:
- [Result] Negi S, Shukrullah I, Veledar E, Bloom HL, Jones DP, Dudley SC. Statin therapy for the prevention of atrial fibrillation trial (SToP AF trial). J Cardiovasc Electrophysiol. 2011 Apr;22(4):414-9. doi: 10.1111/j.1540-8167.2010.01925.x. Epub 2010 Oct 13. PMID 20946227

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Atorvastatin
Started | 31 | 33
Completed | 31 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Atorvastatin | Total
Number analyzed (Participants) | 31 | 33 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (13.9) | 58.2 (11.6) | 58.5 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 26 | 27 | 53

OUTCOME MEASURES:

1. Primary Outcome: Time of Atrial Fibrillation Recurrence
Time Frame: Upon recurrence, up to 12 months
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | Atorvastatin
Number analyzed (Participants) | 31 | 33
days | 22 [7 to 70] | 29 [2 to 145]

2. Secondary Outcome: Comparison of Redox Potential for Cysteine Values
Time Frame: Baseline and 30 days
Measure: Median (Inter-Quartile Range); unit: mV
Arm/Group | Placebo | Atorvastatin
Number analyzed (Participants) | 31 | 33
mV
  Baseline | -61.2 [-71.2 to -54.8] | -65.3 [-71.3 to -58.8]
  1 month (30 day follow-up) | -64.5 [-69.8 to -58.5] | -62.6 [-68.0 to -58.0]

3. Secondary Outcome: Comparison of Redox Potential for Glutathione Values
Time Frame: Baseline and 30 days
Measure: Median (Inter-Quartile Range); unit: mV
Arm/Group | Placebo | Atorvastatin
Number analyzed (Participants) | 31 | 33
mV
  Baseline | -116.7 [-134.9 to -110.2] | -125.3 [-138.0 to -117.3]
  1 month (30 day follow-up) | -124.3 [-142.1 to -109.0] | -129.0 [-138.2 to -113.4]

4. Secondary Outcome: Comparison of Derivatives of Reactive Oxygen Metabolites Values
Time Frame: Baseline and 30 days
Measure: Median (Inter-Quartile Range); unit: Carr
Arm/Group | Placebo | Atorvastatin
Number analyzed (Participants) | 31 | 33
Carr
  Baseline | 384 [276 to 422] | 382 [322 to 467]
  1 month (30 day follow-up) | 400 [338 to 450] | 345 [304 to 406]

5. Secondary Outcome: Comparison of Isoprostanes Values
Time Frame: Baseline and 30 days
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Placebo | Atorvastatin
Number analyzed (Participants) | 31 | 33
pg/mL
  Baseline | 1259 [1040 to 1738] | 1062 [817 to 1421]
  1 month (30 day follow-up) | 1146 [964 to 1397] | 1240 [953 to 1397]

6. Secondary Outcome: Comparison of Interleukin-6 Values
Time Frame: Baseline and 30 days
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Placebo | Atorvastatin
Number analyzed (Participants) | 31 | 33
ng/mL
  Baseline | 5.3 [2.1 to 9.2] | 4.0 [1.7 to 6.6]
  1 month (30 day follow-up) | 5.6 [3.2 to 8.6] | 2.2 [1.7 to 3.6]

7. Secondary Outcome: Comparison of Interleukin-1 Values
Time Frame: Baseline and 30 days
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Placebo | Atorvastatin
Number analyzed (Participants) | 31 | 33
ng/mL
  Baseline | 0.29 [0.20 to 0.44] | 0.30 [0.17 to 0.47]
  1 month (30 day follow-up) | 0.25 [0.17 to 0.32] | 0.28 [0.21 to 0.32]

8. Secondary Outcome: Comparison of High Sensitivity C-reactive Protein
Time Frame: Baseline and 30 days
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Placebo | Atorvastatin
Number analyzed (Participants) | 31 | 33
mg/L
  Baseline | 9.6 [1.7 to 15.0] | 6.3 [2.2 to 11.8]
  1 month (30 day follow-up) | 12.3 [2.8 to 14.4] | 2.3 [1.3 to 4.7]

9. Secondary Outcome: Comparison of Tumor Necrosis Factor Alpha Values
Time Frame: Baseline and 30 days
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Placebo | Atorvastatin
Number analyzed (Participants) | 31 | 33
ng/mL
  Baseline | 2.0 [1.2 to 2.9] | 1.8 [1.4 to 2.5]
  1 month (30 day follow-up) | 2.6 [1.7 to 3.8] | 1.5 [1.2 to 2.9]

ADVERSE EVENTS:
Arm/Group | Placebo | Atorvastatin
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/33
Other Adverse Events (participants affected / at risk) | 26/31 | 22/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=31) | Atorvastatin (N=33)
Atrial fibrillation (Cardiac disorders) | 26 | 22

LIMITATIONS AND CAVEATS:
Limited enrollment; recurrence rate of AF was slightly higher than other trials indicated that the study sample may be a high-risk population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No